CLINICAL TRIAL: NCT04268290
Title: Effect of Single Incision Plus One Port Laparoscopic Surgery Assistant Enhanced Recovery After Surgery on Colorectal Cancer : A Single Arm Trial
Brief Title: Single Incision Plus One Port Laparoscopic Surgery Assistant Enhanced Recovery After Surgery on Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2019-156
Record Dates: First submitted 2019-12-25; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; ERAS; Single Incision plus one; Laparoscopic surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SILS plus one assistant ERAS (Experimental): Preoperative:
  preadmission information, education, counseling, optimization ( breathing training), shortening fasting time and carbohydrate load
  Intraoperative:
  The intravenous fluid therapy is restricted. All patients undergo single incision plus one port laparoscopic surgery(SILS plus one).
  A suitable warming device (such as forced-air heating blankets) and warmed intravenous fluids are been adopted routinely to keep body temperature
  Postoperative:
  multimodal analgesia (surgical site infiltration, a nonsteroidal anti-inflammatory drug, epidural analgesia) early oral intake and move. nasogastric tubes should not be used routinely. Nasogastric tubes inserted during surgery are been removed before reversal of an aesthesia.
  Interventions: Combination Product: Single incision plus one port laparoscopic surgery

INTERVENTIONS:
Combination Product: Single incision plus one port laparoscopic surgery — SILS plus one port surgery and enhanced recovery after surgery protocol both are methods taking the minimally invasive benefits for the patients including faster recovery, reduced postoperative pain and shorter hospital stay.
  Other Names: The program of enhanced recovery After Surgery

SUMMARY:
Conventional laparoscopic surgery (CLS) for colorectal cancer has been demonstrated to be safe and feasible and present minimally invasive benefits including faster recovery, reduced postoperative pain and shorter hospital stay, also acquiring comparable oncologic outcomes with open surgery. To achieve further minimally invasive outcomes, SILS plus one port surgery was attempted by some surgeons. Preliminary results showed that SILS+1 could achieve better minimally invasive benefits than CLS while preserving oncologic feasibility.

Till now, ERAS has been practiced in colorectal cancer surgery for approximately 20 years. Studies have proven that ERAS is safe and significantly improved the recovery course of patients during perioperative period, meanwhile, the expense could be greatly reduced.

Based on ERAS studies protocols and SILS+1 trials, investigators tried to combine SILS+1 with ERAS, hopefully to provide patients with more safe, economic, feasible and rapid surgery and perioperative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Primary tumor diagnosed as adenocarcinoma confirmed pathologically by endoscopic biopsy
* cT1-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition
* Located in the cecum, ascending colon, transverse colon, descending colon, sigmoid colon, the upper segment of the rectum.
* Diameter ≦ 5cm
* No severe organ dysfunction
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I or II
* Written informed consent

Exclusion Criteria:

* Unsuitable for patients undergoing single incision plus one port laparoscopic surgery
* Patients with Complications caused by colorectal cancer ( bleeding , perforation, obstruction or incomplete obstruction )
* Previous abdominal surgery
* Malignant diseases within the past 5years
* Requirements of simultaneous surgery for another diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Rehabilitative rate | 4 days
  The percentage of patients who met discharge criteria in the fourth day after surgery
Postoperative hospital stays | 1 month
  Days from surgery to discharge

SECONDARY OUTCOMES:
Medical cost | 1 month
  The patient's expenses from surgery to discharge are recorded in RMB "yuan"
Postoperative pain score | Once a day from 6 hours to the fourth day after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score tool on postoperative day . On a scale of 1 to 10, the higher the score, the greater the pain.
Postoperative recovery index | 1 month
  The first Time to early mobilization(hour), flatus(hour), liquid diet(hour), soft diet(hour), removal of the Nasogastric tubes(hour) , removal of the peritoneal drainage(hour) are used to assess the postoperative recovery
Postoperative inflammatory immune response | 3 days
  It includes the number of white blood cells and lymphocytes,CRP, IL-6
compliance with ERAS measures | perioperative
  It is defined as if the patients complete every ERAS measure or not. We can defined it "yes " or "not".
6 min postoperative walking test(6MWT) | Once a day from the frist to the fourth day after surgery
  Study site, subject preparation, trial procedures, and medical monitoring refer to the 6MWT guidelines issued by the American thoracic society in 2002.
hospital readmissions | 30days
  It can be defined as the number of patients readmitted within 30 days because of postoperative complications.
Morbidity and mortality rates | 30 days
  Morbidity and mortality rates are defined as postoperative complications graded according to Clavien-Dindo within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yannan, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Derived] Zhang X, Li G, Li X, Liang Z, Lan X, Mou T, Xu Z, Fu J, Wu M, Li G, Wang Y. Effect of single-incision plus one port laparoscopic surgery assisted with enhanced recovery after surgery on colorectal cancer: study protocol for a single-arm trial. Transl Cancer Res. 2021 Dec;10(12):5443-5453. doi: 10.21037/tcr-21-1361. PMID 35116390